CLINICAL TRIAL: NCT01196962
Title: A Randomize Controlled Trial to Compare the Complications of Subclavian and Internal Jugular Venous Catheterization in Critically Ill Patients
Brief Title: Safety Study of Subclavian and Internal Jugular Venous Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSIS; EDAH (Other: EDAH)
Record Dates: First submitted 2010-09-01; First posted 2010-09-09 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2011-08

CONDITIONS: Time to Insertion; Rates of Complications
Keywords: central venous catheter; complications; internal jugular vein; randomized trial; subclavian vein
MeSH Terms: interventions — Central Venous Catheters; Vascular Access Devices

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Internal jugular vein (Experimental)
  Interventions: Device: Central venous catheter

INTERVENTIONS:
Device: Central venous catheter — Central venous catheter insertion to subclavian vein
  Other Names: venous access

SUMMARY:
There is no randomized controlled trial to compare the rates of complications associated with internal jugular and subclavian venous catheterization. The aim of this study is to compare mechanical, infectious, and thrombotic complications of internal jugular and subclavian venous catheterization. An improved understanding of CVC-related risks might help clinicians to choose one approach over the other in specific clinical settings.

DETAILED DESCRIPTION:
Central venous catheterization is often necessary to treat critically ill patients hospitalized in intensive care units (ICUs). However, this procedure may lead to serious and sometimes life-threatening complications, including mechanical, infectious, or thrombotic complications. The choice of insertion site can influence the incidence and type of such complications. The most frequently used sites for CVC insertion are the internal jugular and the subclavian vein. However, in an individual patient, criteria for choosing one approach over the other remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* admission to ICU
* requiring central venous catheterization
* without contraindications to attempt both jugular and internal jugular access

Exclusion Criteria:

* the presence of a central venous catheter at admission
* central venous catheterization within 2 weeks prior to admission
* emergency catheterization for a life-threatening situation
* major blood coagulation disorders
* anatomic defect precluding catheterization at either site
* skin lesions or recent surgery at either site

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Time to completely insertion | 1 hour

SECONDARY OUTCOMES:
rates of mechanical, infectious, and thrombotic complications | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Feng Wei, M.D., Principal Investigator — Chest department
Locations (1):
- E-Da hospital, Kaohsiung City, Taiwan